CLINICAL TRIAL: NCT01804777
Title: ENaC as a Novel Mechanism for Hypertension and Volume Expansion in Type 2 Diabetes
Brief Title: Epithelial Sodium Channel (ENaC) as a Novel Mechanism for Hypertension and Volume Expansion in Type 2 Diabetes
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Currently closed for data analysis.
Sponsor: University of New Mexico (Other)
Collaborators: Dialysis Clinic, Inc. (Industry); University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: 13-017
Record Dates: First submitted 2013-03-01; First posted 2013-03-05 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Proteinuria; Hypertension; Type II Diabetes
Keywords: ENaC; Amiloride; Hydrochlorothiazide(HCTZ); Hypertension; Type II Diabetes; Natriuresis; Proteinuria
MeSH Terms: conditions — Proteinuria; Hypertension; Diabetes Mellitus, Type 2 | interventions — Amiloride; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amiloride 10 mg, 20 mg, and diet (Experimental): Amiloride 10 mg for 14 days and diet. Then dose titrated up at day 14 to 20 mg, and diet.
  Interventions: Drug: Amiloride
- HCTZ 12.5 mg, 25 mg and diet (Active Comparator): HCTZ 12.5 mg for 14 days and diet. Then dose titrated up at day 14 to 25 mg, and diet
  Interventions: Drug: HCTZ

INTERVENTIONS:
Drug: Amiloride — Amiloride 10 mg taken every day for two weeks, along with adherence to specified diet.
  On day 14 titrate dose up to Amiloride 20 mg, take every day for two weeks after completion of two week intake of Amiloride 10 mg, along with adherence to specified diet.
  Other Names: Midamor
  Arms: Amiloride 10 mg, 20 mg, and diet
Drug: HCTZ — HCTZ 12.5 mg taken every day for two weeks, along with adherence to specified diet.
  On day 14 titrate dose up to HCTZ 25 mg taken every day for two weeks after completion of two week intake of HCTZ 12.5 mg, along with adherence to specified diet
  Other Names: Hydrochlorthiazide; Aquazide H; HydroDIURIL; Microzide
  Arms: HCTZ 12.5 mg, 25 mg and diet

SUMMARY:
The purpose of this study is to determine with the administration of amiloride, observe an enhanced natriuresis, reduction in blood pressure and weight compared to the administration of hydrochlorothiazide in Type 2 Diabetics.

DETAILED DESCRIPTION:
Renal sodium retention and extracellular fluid volume expansion are hallmarks of nephrotic syndrome. There is abundant evidence that this occurs even in the absence of activation of hormones that are known to activate renal Na transporters. Proteinuria not only reflects glomerular damage, but also functions as a risk factor for cardiovascular disease, stroke, end stage renal disease and is associated with extracellular volume expansion and high BP.

In the natural course of Type II diabetes, microalbuminuria and elevations in blood pressure are thought to occur at around the same time. Blood pressure in microalbuminuric diabetics is more sensitive to dietary salt intake than in normoalbuminuric patients despite both groups having similar aldosterone and plasma renin activity levels. Proteolytic processing of ENaC subunits might provide the primary defect in renal sodium handling in these microalbuminuric individuals. However, proteinuria is not consistently identified as a risk factor for incipient elevation in blood pressure and in some studies elevated blood pressure predicts the advent of microalbuminuria.

Analyses of normotensive normoalbuminuric subjects in previous studies have found that higher urinary albumin levels in the normal range predicted incident hypertension. A similar finding was seen in a non-diabetic cohort. These studies suggest that these disparate results may be related to the cut off that defined microalbuminuria. Another possible explanation is that an ENaC activator, like plasmin, contributes to the generation of incident hypertension in some individuals. Levels of albuminuria may not necessarily be reflective of ENaC activator levels and may vary from individual to individual. Perhaps urinary plasmin and plasminogen provides a more robust biomarker for those individuals who may develop hypertension.

Recent evidence suggests that in some individuals with glomerular damage, proteases not normally found in urine enter the urinary space and aberrantly cleave ENaC. In this setting, filtered plasminogen (inactive precursor) is converted to plasmin (active protease) by urokinase that is expressed in tubular epithelial lumen. The proteolytic activation of ENaC would generate a primary defect in renal sodium handling, a mechanism that may be a particularly important factor leading to increases in extracellular fluid volume and BP that accompany nephrotic syndrome.

While previous studies have examined the role of amiloride in low-renin hypertension, and as an additional agent the conventional treatment of hypertension, no human trials have tested whether ENaC inhibitors impact blood pressure and volume status in the setting of proteinuria. Over a ten year period, millions of diabetics, 5.3% of Type II diabetics and 28% of Type I diabetics develop macroscopic proteinuria.

ELIGIBILITY:
* Inclusion Criteria:

  1. Age 18 to 80 yrs at randomization
  2. History of Type 2 Diabetes
  3. Presence of systolic hypertension or pre-hypertension (average systolic blood pressure (SBP) ≥120 mmHg and <180 mmHg.)
  4. Urinary protein/creatinine ratio >300 mg/g creatinine at screening
  5. Hemoglobin A1C<8%
  6. Willing and able to give informed consent
* Exclusion Criteria:

  1. Average SBP of ≥180 mmHg or diastolic blood pressure (DBP) of ≥110 mmHg
  2. Current symptomatic heart failure, history of New York Heart Association Class III or IV congestive heart failure, or left ventricular (LV) ejection fraction (by any method) <25%; these patients may be harmed with withdrawal of diuretics
  3. Serum potassium level <3.5 or >5.0 at screening
  4. History of hyperkalemia in the last two years (serum K>5.5)
  5. Contraindication to use of hydrochlorothiazide or amiloride
  6. Unstable angina pectoris or acute myocardial infarction (MI) in last 3 months
  7. Known secondary causes of hypertension (HTN) (screening for these conditions will not be required)
  8. Estimated glomerular filtration rate (GFR) <60 mL/min/1.73m², as determined by validated estimating equations
  9. On or expected to be on immunosuppressive therapy
  10. Any history of solid organ transplantation
  11. Significant dementia
  12. Other factors likely to limit adherence during trial (eg. alcohol or substance abuse, plan to move in next year, history of non-adherence to medications, appointments and medical care, reluctance of close family members to participate in trial, lack of support from primary healthcare provider)
  13. Participation in another investigational trial within 4 weeks of the screening visit
  14. Arm Circumference too large or too small to allow accurate blood pressure measurement
  15. Pregnancy or currently trying to become pregnant (although this is unlikely because of age limit
  16. Incarceration

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | one month
  Change in clinic systolic BP. This BP measure will be the average of three serial BP measurements taken one minute apart after 5 minutes of sitting quietly.

SECONDARY OUTCOMES:
Hypertension | one month
  To demonstrate effect size on relevant hypertension outcomes such as volume status and urinary sodium excretion. Also assess the fractional excretion of sodium (FENa) and chloride (FECI). Endpoint will be the 24 hour urine excretion.

CONTACTS AND LOCATIONS:
Overall Officials: Mark L Unruh, MD MSc, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico Hospital; Clinical & Translational Science Center, Albuquerque, New Mexico, United States

REFERENCES:
- [Background] Passero CJ, Hughey RP, Kleyman TR. New role for plasmin in sodium homeostasis. Curr Opin Nephrol Hypertens. 2010 Jan;19(1):13-9. doi: 10.1097/MNH.0b013e3283330fb2. PMID 19864949